CLINICAL TRIAL: NCT03079596
Title: Comparison of ERAS (Early Recovery After Surgery) Protocol With Conventional Protocol After Laparoscopic Total Gastrectomy and Proximal Gastrectomy: A Prospective Randomized Controlled Trial (Phase II Study)
Brief Title: ERAS (Early Recovery After Surgery) Protocol After Laparoscopic Total Gastrectomy and Proximal Gastrectomy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Seoul National University Bundang Hospital (Other)
Responsible Party: Principal Investigator, Sang-Hoon Ahn, Profesor, Seoul National University Bundang Hospital
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: B-1608-357-006
Record Dates: First submitted 2017-03-09; First posted 2017-03-14 (Actual); Last update posted 2021-08-11 (Actual); Status verified 2021-08

CONDITIONS: Gastric Cancer
Keywords: gastric cancer; ERAS (early recovery after surgery); laparoscopic total gastrectomy
MeSH Terms: conditions — Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- ERAS perioperative cares (Active Comparator): Patients planned to undergoing laparoscopic total gastrectomy, following the ERAS protocols
  Interventions: Procedure: ERAS perioperative cares
- Conventional perioperative cares (Active Comparator): Patents will be managed by our hospital's critical pathways
  Interventions: Procedure: Conventional perioperative cares

INTERVENTIONS:
Procedure: ERAS perioperative cares — Patient's preoperative counseling & education before surgery No Bowel preparation Oral Carbohydrate Solution (OCS) loading until 2hours before surgery Fluid restriction & Management by pulse contour analysis or transesophageal doppler Early mobilization Early oral feeding (postoperative 1 day - sips of water, 2 days - semifluid diet (SFD), 3 days - soft blended diet (SBD)) Epidural patient controlled analgesics (no opioids analgesics) Postoperative Nausea Active Control Thromboembolism prophylaxis by low molecular weighted heparin (LMWH) Perioperative High content Oxygen therapy No drain insertion No Levin tube Patients will be discharged at POD#4 if there's no problem.
  Arms: ERAS perioperative cares
Procedure: Conventional perioperative cares — No Patient's preoperative counseling & education before surgery Bowel preparation No Oral Carbohydrate Solution (OCS) loading until 2hours before surgery Conventional Fluid Management by clinical signs (Urine output, heart rate etc.) Conventional Mobilization Conventional oral feeding (POD#2 SOW, #3 SFD, #4 SBD) IV PCA Postoperative Nausea Control if needed No Thromboembolism prophylaxis No or Low Content Oxygen therapy Routine drain insertion Levin tube insertion if needed
  Arms: Conventional perioperative cares

SUMMARY:
Enhanced Recovery After Surgery (ERAS) programs have been introduced with purposes of reducing the surgical stress response and obtaining optimal recovery after surgery.

DETAILED DESCRIPTION:
There is strong evidence of the usefulness of the ERAS programs in patients undergoing colorectal surgery in terms of significantly reduced postoperative complications and shorter length of hospital stay, compared to the patients of conventional treatment.

However, few studies exist about the implication of ERAS programs in the laparoscopic gastrectomy.

The aim of this study was to compare the recovery rate, morbidity, and quality of life in the patients undergoing laparoscopic total gastrectomy and proximal gastrectomy for gastric cancer, receiving either ERAS protocol or conventional postoperative cares.

ELIGIBILITY:
Inclusion Criteria:

* Elective surgery
* American Society of Anesthesiologists (ASA) scores < 3
* Gastric cancer, adenocarcinoma, possible to perform laparoscopic total gastrectomy and proximal gastrectomy
* Informed consent
* No other treatment (Radiation, Chemotherapy or Immunotherapy) on this gastric cancer or other type of cancer.
* No systemic inflammatory disease

Exclusion Criteria:

* conversion to open

Ages: 20 Years to 68 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2019-10-01 (Actual); Primary Completion 2022-10-01 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Tolerance of diet for 24 hours | 4 days after surgery
  Tolerance of diet for 24 hours. Able to eat one third of more of soft-blend meal without abdominal discomfort, bloating, nausea, or vomiting
Analgesic-free | 4 days after surgery
  Analgesic-free (oral or IV analgesic drugs not necessary after cessation of PCA)
Safe ambulation | 4 days after surgery
  Safe ambulation (ambulation of 600m without assistance)
Afebrile status without major complications | 4 days after surgery
  Afebrile status without major complications (fever defined as body temperature greater than 37.5)

SECONDARY OUTCOMES:
Postoperative length of hospital stay | up to 4 weeks after surgery
  Postoperative length of hospital stay
Time to tolerance of a full diet | up to 1 month after surgery
  Time to tolerance of a full diet
Time to first bowel motion | up to 7 days after surgery
  Time to first bowel motion

CONTACTS AND LOCATIONS:
Locations (1):
- Seoul National University Bundang Hospital, Seongnam-si, Gyeonggi-do, South Korea

IPD SHARING:
Plan to Share IPD: No